CLINICAL TRIAL: NCT06125587
Title: Chiglitazar Versus Metformin for Insulin Resistance in Non-obese Patients With Polycystic Ovary Syndrome
Brief Title: Chiglitazar/Metformin in Non-obese Women With PCOS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yining Yang, Principal Investigator, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023PS581K
Record Dates: First submitted 2023-11-05; First posted 2023-11-09 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Polycystic Ovary Syndrome; Chiglitazar; Metformin
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — chiglitazar; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chiglitazar group (Experimental): Chiglitazar, tablet, 32mg, taken orally once daily for 3 months
  Interventions: Drug: Chiglitazar
- Metformin group (Active Comparator): Metformin, tablet, 0.5g, taken orally twice daily for 3 months
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Chiglitazar — Chiglitazar is a novel PPAR agonist. Treatment of type 2 diabetes mellitus by moderate activation of PPARα, PPARγ and PPARδ, improving insulin sensitivity, regulating blood glucose, and promoting fatty acid oxidation and utilization.
  Arms: Chiglitazar group
Drug: Metformin — Metformin is not only an antihyperglycemic drug, it also corrects insulin resistance and hyperandrogenism in polycystic ovary syndrome.
  Arms: Metformin group

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common endocrine and metabolic disorders in women of reproductive age, and its prevalence rate is from 9% (NIH criteria) to 18% (Rotterdamcriteria). It is clinically characterized by hyperandrogenism, persistent anovulation, and polycystic ovarian changes. Moreover it is often accompanied by insulin resistance and obesity. Now, metformin is not only an antihyperglycemic drug, it also corrects insulin resistance and hyperandrogenism in polycystic ovary syndrome. Chiglitazar is a novel peroxisome proliferation activated receptor (PPAR) agonist. Treatment of type 2 diabetes mellitus by moderate activation of PPARα, PPARγ and PPARδ, improving insulin sensitivity, regulating blood glucose, and promoting fatty acid oxidation and utilization. However, there is limited evidence for its treatment of insulin resistance in women with PCOS. Therefore, investigators applied chiglitazar and metformin to two groups of PCOS patients to understand their effects on insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 18- 45 years old
2. Normal weight BMI 18.5--24
3. Diagnosis of hyperandrogenism T>0.481ng/ml
4. The diagnosis of PCOS is based on the diagnostic criteria established by the Rotterdam consensus
5. No use of drugs affecting reproductive endocrine in the 3 months prior to the clinic visit

Exclusion Criteria:

1. T level is within the normal range
2. Organ dysfunction
3. Drugs that can affect endocrine such as contraceptives and steroids taken in the past 3 months
4. Confirmed diagnosis of diabetes
5. Are on a diet, use weight-affecting medications, or have experienced a weight change of >4.5kg within 3 months prior to the start of the study
6. Have other endocrine disorders, such as thyroid dysfunction, adrenal gland disease, hyperprolactinemia, etc.
7. Combined psychiatric disorders and severe primary diseases
8. Allergy to the drug or components of this study
9. Those who do not follow the doctor's instructions during the medication, or discontinue the treatment due to serious adverse reactions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Plasma insulin level | Three months
  Changes in insulin level before and after treatment

SECONDARY OUTCOMES:
Total testosterone | Three months
  Changes in total testosterone (TT)
Sex hormone-binding globulin | Three months
  Changes in sex hormone-binding globulin (SHBG)
Ratio of luteinizing hormone to follicular estrogen | Three months
  Changes in ratio of luteinizing hormone to follicular estrogen (LH/FSH)
BMI and WHtR | At baseline and at 12 weeks after randomization via a standardized protocol.
  Anthropometric indices, including height, weight, waist-to-height ratio (WHtR) and BMI, were assessed at baseline and at 12 weeks after randomization via a standardized protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang Y, Han Y, Xu J, Gao Y, He B. The effects of chiglitazar and metformin on insulin resistance in women with a normal BMI and polycystic ovary syndrome: a randomized controlled study. BMC Endocr Disord. 2025 Dec 2;25(1):283. doi: 10.1186/s12902-025-02082-0. PMID 41331576